CLINICAL TRIAL: NCT05701787
Title: Molecular Landscape Analysis and Clinical and Therapeutic Implications for NSCLC Patients With Rare Mutations
Brief Title: Molecular Landscape Analysis and Clinical Implications for NSCLC Patients With Rare Mutations
Status: Recruiting | Type: Observational
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xiaomin Niu, Principal Investigator, Shanghai Chest Hospital
Other Study IDs: THORACIC003
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-04

CONDITIONS: NSCLC; NSCLC Stage IV; NSCLC, Recurrent
Keywords: NSCLC; rare mutations; molecular landscape; next-generation sequencing (NGS); targeted therapy; immunotherapy; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lung cancer is the most common primary cancer of the lung and is responsible for the ever increasing number of cancer-related deaths worldwide. Especially in China, the burden of lung cancer has been rising rapidly due to its large and growing population. Histologically, approximately 85% of lung cancers are non-small-cell lung cancer (NSCLC).

Molecular targeted therapy has been shown to dramatically improve the quality of life and survival outcomes of NSCLC patients. One of the most important targeted drugs in NSCLC has been the epidermal growth factor receptor-tyrosine kinase inhibitors (EGFR-TKIs), while there exists some other rare targetable mutation in NSCLC. Emerging evidence underlines that, rather than a single point mutation, some rare mutations present with a wide array of mutations, essentially in NSCLC.

Different rare mutations with NSCLC have divergent clinical and therapeutic implications with a particular distinction. Therefore, there is an unmet need for more effective therapies for NSCLC with rare mutations. In summary, identification of genetic alterations in NSCLC with rare mutations is increasingly essential to perform molecular diagnostics and individualized treatments. This project aims to create a registry of patients with NSCLC with rare mutations to further the characterization of molecular alterations and develop (novel) treatments based on the detection.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of NSCLC with rare mutations including EGFR rare mutations, ALK fusion, ROS1 fusion, BRAF V600E, cMET exon 14 skipping, KRAS G12C, RET fusion, NTRK fusion, etc.
* 18 years of age or older
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants with NSCLC with rare mutations are with the standard treatment and/or are enrolled in the clinical trials.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 20 years
  Collect detailed clinical information on patients with NSCLC with rare mutations via the electronic medical records
Disease control rate (DCR) | 20 years
  Collect detailed clinical information on patients with NSCLC with rare mutations via the electronic medical records
Progression-free survival (PFS) | 20 years
  Collect detailed clinical information on patients with NSCLC with rare mutations via the electronic medical records

SECONDARY OUTCOMES:
Overall survival (OS) | 20 years
  Collect detailed clinical information on patients with NSCLC with rare mutations via the electronic medical records

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomin Niu, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Xiaomin Niu, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No